CLINICAL TRIAL: NCT06868524
Title: Leveraging Adaptation and Multilevel Implementation Strategies to Address Unique Health Promotion Challenges Among Cancer Survivors
Brief Title: Leading Healthy Eating and Activity Promotion Program
Acronym: LEAP
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300010921; 1U54CA280770-01 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cancer Survivor; Cancer; Oncology
Keywords: cancer survivor; cancer; oncology; exercise; nutrition; diet; healthy lifestyle; behavior change
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Program participants: Agree to evaluate a community-based, publicly available program combining a website with optional in person group sessions.

SUMMARY:
The goal of the LEAP project is to improve the health and well-being of cancer survivors and their co-survivors living in persistent poverty areas by providing healthy behavior change support. This will be done by engaging the community in adapting beneficial approaches for promoting healthy diet and regular physical activity into a program for cancer survivors and co-survivors that is appropriate for the persistent poverty context and social determinants of health.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 89
* English speaking
* Resident of Birmingham area or surrounding community
* History of any type of cancer or the friend or family with of a cancer survivor

Exclusion Criteria:

* Serious difficulty hearing
* History of dementia or organic brain syndrome
* On primary treatment for cancer
* No other other medical, psychological, or social characteristic that would interfere with participation in evaluation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cancer survivors or the friend/family member of a cancer survivor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that meet the dietary guidelines for healthy diet | Baseline, 12-weeks
  Measuring the number of participants that meet the dietary guideline's recommendations for fruit and vegetable intake and added sugar.
Number of participants that meet the recommended minutes of physical activity per week | Baseline, 12-weeks
  Measuring physical activity from one-week of wearing an accelerometer
Overall quality of life score | Baseline, 12-weeks
  self reported survey to collect data about physical, mental, and social health on a scale of 1 to 5 with 5 being excellent and 1 being poor
Change in BMI | Baseline, 12-weeks
  Trained research staff will measure height using portable stadiometer (baseline only; no shoes) and weight using portable calibrated scale (light clothing without shoes) to calculate BMI (weight in kg/height in meters squared)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Rogers, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individuals interested in requesting IPD should contact the study PIs.
Supporting Information: ICF
Time Frame: After data management is finalized (and data locked) and the main outcomes manuscript has been submitted.
Access Criteria: A data use agreement between the institution housing the data (UAB) and the institution of the requesting researcher will be required.